CLINICAL TRIAL: NCT03377088
Title: Aromatherapy for Management of Back Pain in the Emergency Department
Brief Title: Aromatherapy Randomization of Pain Management in Adults
Acronym: AROMA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Principal Investigator and Vice Chair of EM Research, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1116889-3
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Back Pain; Back Pain, Low; Sciatica
MeSH Terms: conditions — Back Pain; Low Back Pain; Sciatica | interventions — Oils, Volatile; almond oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond Oil (Placebo Comparator): Patients will be given Almond Oil for inhalation on cotton balls as a control. Almond Oil has been shown to act as a placebo when compared to our variable, Rosa Damascena oil. To ensure blinding, this arm will act to always deliver a scent to a patient, blinding them to whether they are receiving a known aromatherapy or a common scent.
  Interventions: Other: Almond Oil
- Rose Oil (Experimental): Patients will be given Rosa Damascena oil on cottons balls as a variable. This oil has been shown to significantly lower acute pain levels on the visual analog pain scale when compared to placebo of distilled water or Almond Oil.
  Interventions: Other: Rose oil

INTERVENTIONS:
Other: Rose oil — Rose oil will be given as the intervention in this study, an over-the-counter agent that can be commonly found in retail stores. It will be delivered as 2 drops 50% rose oil in water on a cotton ball within 20 cm of the patient's face for 30 minutes.
  Other Names: Rosa Damascena (Damask Rose) essential oil
  Arms: Rose Oil
Other: Almond Oil — Almond Oil has been shown in limited studies to act as a placebo for pain control when compared to Rose Oil. This subtly sweet oil will be used to ensure the patient always receives a smell, and maintains blinding.
  Other Names: Sweet almond oil
  Arms: Almond Oil

SUMMARY:
Pain control for acute isolated back pain and sciatica is a nebulous and often illusive task in the emergency department, and a challenge face everyday by emergency medicine physicians. Standard pain control practices are poorly defined in practice and in the literature. NSAIDs alone have been shown to be less-than-adequate controllers of acute back pain warranting emergency department visits and have little bearing on long-term pain control or recovery. Opioids are additionally poor long-term pain controllers and are gaining public controversy for their overuse. Modalities such as acupuncture, massage, thermotherapy, and spinal manipulation have been described in the literature with minimal evidence. Aromatherapy for pain control has been recently demonstrated as effective in the management of burn-dressing changes as well as post-operative pain management in children. It is an inexpensive and easily employed modality not yet explored in the emergency department for acute pain such as isolated back pain and sciatica. The authors propose to study Rosa damascena oil aromatherapy for the control of isolated acute back pain in the emergency department compared to almond oil placebo. The authors hypothesize that Rosa damascena will provide additional pain relief, as a known analgesic, when compared to almond oil aromatherapy. The authors will identify patients presenting to the Stony Brook University Hospital (SBUH) Emergency Department (ED) with acute isolated back pain and sciatica and test this hypothesis using a blind randomized approach. Patients included will be those above the age of 18 with isolated, non-traumatic back pain and sciatica lasting less than 2 weeks. Primary outcomes measured will include decrease in pain severity on a visual analog scale after 30 minutes of aromatherapy and again at 60 minutes post-therapy. Secondary outcomes measured will include patient satisfaction, need for clinician-determined rescue medications, and minimal clinical importance difference of pain control. Aromatherapy will be provided with both essential oil concentrated Rosa damascena and almond extract delivered via soaked-cotton ball 20-30 cm from the patient's face.

DETAILED DESCRIPTION:
A. SPECIFIC AIMS This study aims to research the use of aromatherapy for pain control in the emergency department, specifically, acute back pain. Aromatherapy, particularly Rose Essential Oil (Rosa damascena) has been studied in recent literature and shown to be effective versus placebos for the control of acute pain with lasting effects during burn dressing changes and post-operative pain management. These studies have been small and specific to discrete clinical conditions. Their evidence supports the use of aromatherapy for acute pain control with additional patient satisfaction benefit, but they are not yet externally validated to more common conditions facing emergency medicine physicians. The investigators chose to study acute isolated back pain and sciatica presenting to the emergency department and the use of Rosa damascena essential oil versus a control of Almond Oil for the treatment of isolated back pain and sciatica. The authors will investigate the use of aromatherapy in pain management by measuring and comparing pre- and post-treatment pain levels using a 100 mm visual analog scale (VAS) for pain. A significant reduction in pain by 13 mm on the VAS has been previously demonstrated as the minimal clinically important difference for treatment of pain. The primary endpoint will be the evaluation of significant change in VAS score greater than 13 mm between both groups immediately following a 30 minute blinded aromatherapy treatment and again 30 minutes later. The secondary endpoints include patient satisfaction, need to rescue medication (its type and dose), and subjective changes in pain.

B. Background and Significance Aromatherapy has been hypothesized to be an effective management strategy for acute pain control. Its use has been recently demonstrated in Iran, using Rosa damascena (Damask Rose) essential oil. Rosa damascena is believed to possess anti-anxiolytic, sedative, anticonvulsive, and analgesic effect on the central nervous system (CNS) when delivered through the olfactory system (Mohebitabar et al. 2016). This theory is believed to be in part due to the lateral gate theory of pain control and a stimulant's ability to inhibit transmission of stimuli through pain fibers. However, while any olfactory stimulant might be hypothesized to do just that, only Rosa damascena has been shown to produce significant reduction in pain on the VAS as well as patient satisfaction when compared to scented placebos like Almond Oil. Rosa damascena has been shown to improve pain control during dressing changes of second- and third-degree burns (Bikmoradi et al 2016). It has also been shown effective and equal to NSAID treatment of immediate post-operative pain in children (Marofi et al. 2015). It may be an affordable and easy-to-use modality for pain control in the emergency department. Its prior studies are small in sample size and carry little external validity that could be applied to an American Emergency Department population. The authors aim to assess whether aromatherapy using Rosa Damascena is reproducible in the emergency department for control of isolated and acute back pain, two common painful conditions seen with poor evidence for proper pain control. Validity of Rosa damascena aromatherapy in acute back pain and sciatica may open new doors of pain control to be researched in the emergency department and will further characterize the use of aromatherapy in modern medicine.

C. Preliminary Studies The known external studies of Rosa damascena have been cited above and will be presented in the references section. The authors have not yet studied aromatherapy in the emergency department and will be completing this study fresh, based on methodology used in external aromatherapy and back pain treatment studies. The Minimal Clinically Important Difference (MCID) of 13 mm on the VAS has been studied repeatedly and validated as the minimal VAS change needed for a patient to express significantly subjective improvements in pain (Gallagher, Leibman, and Bijur 2001)(Jensen and Chen 2003). Successful pain treatment has been shown by using 3-5 drops of 40% Rosa damascena oil on a cotton ball or gauze pad 20-30 cm from a patients face for 30 minutes (Bikmoradi et al. 2016). Additionally, uses of rescue medications and patient satisfaction have been commonly used as secondary measures in both aromatherapy and landmark back pain treatment studies. Patient demographics include age, gender, comorbidities, prior treatment, BMI, education, marital status, and pain identifiers have been repeatedly used to assess patient demographic distribution in many benchmark Emergency Medicine acute pain management studies (Chang et al 2015.)(Friedman et al. 2015).

D. Research Design and Methods

Rationale and Overview Isolated acute back pain (less than 2 weeks duration) and sciatica are common complaints to the emergency department requiring acute pain management with often chronic follow-up. Their abundance in the ED as well as poorly defined treatment recommendations make them an excellent candidate to study the use of aromatherapy in the emergency department. The authors will replicate the Rosa damascena trials referenced above in similar protocols, patients will be recruited if they fit the attached inclusion criteria and do not meet exclusion criteria. Patients will be treated with either Almond Oil extract or Rosa damascena extract, and both the investigator and patient will be blinded to the control arm. A VAS pain scale will be recorded before treatment, after 30 minutes of treatment, and after a following 2nd 30 minutes. Patients will additionally be asked about their satisfaction and subjective changes in pain, they will be blinded to their prior VAS line placements for proper evaluation of objective pain level changes. Demographics thought to contribute to the sensation of pain, expression of pain, and response to pain treatment will additionally be collected without entangling Private Health Information (PHI). Finally, the use of rescue medication such as NSAIDs or Narcotics at the treating physician's discretion will be recorded as an indicator of treatment failure and complication. Pain will be qualified in its type, locations, duration, immediate episodes prior to presentation, and prior remote episodes in the patient's lifetime health history. Pain will also be quantified by attempted at-home treatments prior to presentation.

Research Site The entirety of this prospective clinical trial will be conducted at the Stony Brook Hospital Emergency Department, an ED with over 110,000 annual visits.

Study Sample Patients will be recruited into this study by an investigator in the Stony Brook Emergency Department. A sample size was calculated to be 30 patients for each treatment arm based on a power of 0.80, desired p value below 0.05, and 95% confidence intervals with the anticipated possibility of patient loss or desire to withdraw during treatment. Patients will be approached for recruitment after an attending or resident physician has seen them and does not anticipate immediate need for narcotic pain medication, immediate imaging, or immediate threats to life or limb. Patients will be included by the attached inclusion and exclusion criteria. Double-blinding will be ensured by block randomization of each treatment arm, performed outside of the emergency department. In the Emergency Department Research Offices, the two treatment arms will be allocated into identical, individual vessels with only a codified label applied to each. Using block randomization, 30 treatments will be distributed to each arm in secret by a clinical research assistant or investigator. Each treatment will be codified individually and recorded in secrecy and kept from the investigators. Randomization will then arrange the total 60 treatments in longitudinal order for sequential random treatments to be selected as each patient is recruited.

Screening Patients will be approached in private and the name, title, and role of the investigator explained after asking permission to speak with the patient. The patient will be told that the investigators are conducting a clinical research trial for the treatment of acute back pain and sciatica. Aromatherapy will be explained as the treatment of interest and a modality that has been tested and proven effective in other types of pain. The use of Almond products and Rose products will be briefly discussed with the patients. Patient's will be asked about any allergies and then asked specifically about allergies to Almonds, Roses, perfume, and ibuprofen. Patients will be informed that speaking with the investigator is entirely optional, as is participating in the study, as there may be no direct benefit to them despite disclosure of their private information to the investigator. An Inclusion and Exclusion form will be reviewed with the patient and their chart, noting their sequential patient number in this study as the only de-identified patient ID. No PMI will be collected; no medical record numbers (MRN), address, phone number, emails, name, SSN, DOB, chief complaint, past medical history (PMH), past surgical history (PSH) , or medications will be recorded. The risks and benefits will be explained to the patient including risk of allergy, risk of no change in pain, benefit of pain improvement, and benefit of contribution to medical research. The consent form will be reviewed in full and any questions answered. Those patients interested in participating and able to grant consent will do so.

Procedures Rosa damascena 40% and Almond Oil 40% kept outside of the ED will be prepared each day and dispersed into identical vessels with randomized identification numbers. The coded numbers and their respective modality will be recorded by an investigator not involved in delivery and kept secured. Patients will be assigned into random treatment arms by block randomization and their coded treatment recorded on the patient data sheet. Patients will be given 4 drops of either modality (40%) on a cotton ball kept between 20 and 30 cm from their face for 30 minutes.

With regards to study blinding, the treatments will be randomly assigned and the patients will not be told which treatment they are receiving. The patients will be aware that the study involves Rose and Almond scents and will likely be able to identify the scent used in their treatment. However, at the end of the study procedures, an independent observer will assess the patient's pain after the aromatherapy has been removed from the room, and will not be aware of which patients received which treatment.

E. Statistics VAS differences immediately after treatment and 30-minutes following will be aggregated from their respective 100 mm VAS for pain and the change calculated for each patient. One-tailed paired t-Tests will be then conducted on the means after standard deviation is calculated and compared between treatment and control groups. A chi-squared test will then be applied between both groups for analysis of significant differences in patient satisfaction and subjective reports of pre- and post-treatment pain. The use of rescue medications by type and dosage will be measured as a percentage of each group and compared via t-Test between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Seen and attending or resident physician
* Isolated back pain or sciatica
* Pain lasting less than 2 weeks
* Pain between lower scapular borders and gluteal folds
* Patient maintains capacity and is interested in participating

Exclusion Criteria:

* Pregnant patient, minor, or inmate patient
* Patient lacks decision making capacity
* Patient is delirious, demented, altered, intoxicated, or agitated
* Patient allergic to Ibuprofen or NSAIDs
* Patient unable to demonstrate understanding of experiment by teach-back method
* Patient below age of 18
* Physician, clinician, or investigator concern for underlying etiology other than isolated back pain or sciatica
* Patient already received narcotics or requires immediate standard pain control
* Patient demonstrated neurologic deficit or radicular symptoms

  * Patient does not wish to be studied
  * Patient endorses allergy to almond, roses, or perfumes
  * Patients with pain lasting greater than 2 weeks

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Acute Pain Reduction | 30 minutes, immediately after treatment
  A 100 mm visual analog scale (VAS) for pain will be administered prior to and after treatment to assess for clinically significant pain control

SECONDARY OUTCOMES:
Patient Satisfaction | 30 minutes (immediately after) treatment
  Patients will be asked after treatment how satisfied they are with their treatment on a 5 point likert scale
Patient Pain Toleration | 30 minutes (immediately after) treatment
  Patients will be asked to subjectively report changes in their pain after completing a VAS pain scale on a 5 point likert scale
Patient Arm Belief | 30 minutes (immediately after treatment)
  Patients will be asked if they think the agent they received was in fact the experimental scent or not, and whether they would consider using it again for future pain control.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital Emergency Department, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Bikmoradi A, Harorani M, Roshanaei G, Moradkhani S, Falahinia GH. The effect of inhalation aromatherapy with damask rose (Rosa damascena) essence on the pain intensity after dressing in patients with burns: A clinical randomized trial. Iran J Nurs Midwifery Res. 2016 May-Jun;21(3):247-54. doi: 10.4103/1735-9066.180380. PMID 27186201
- [Background] Chang AK, Bijur PE, Holden L, Gallagher EJ. Comparative Analgesic Efficacy of Oxycodone/Acetaminophen Versus Hydrocodone/Acetaminophen for Short-term Pain Management in Adults Following ED Discharge. Acad Emerg Med. 2015 Nov;22(11):1254-60. doi: 10.1111/acem.12813. Epub 2015 Oct 19. PMID 26479162
- [Background] Friedman BW, Dym AA, Davitt M, Holden L, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Naproxen With Cyclobenzaprine, Oxycodone/Acetaminophen, or Placebo for Treating Acute Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 20;314(15):1572-80. doi: 10.1001/jama.2015.13043. PMID 26501533
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Marofi M, Sirousfard M, Moeini M, Ghanadi A. Evaluation of the effect of aromatherapy with Rosa damascena Mill. on postoperative pain intensity in hospitalized children in selected hospitals affiliated to Isfahan University of Medical Sciences in 2013: A randomized clinical trial. Iran J Nurs Midwifery Res. 2015 Mar-Apr;20(2):247-54. PMID 25878704
- [Background] Mohebitabar S, Shirazi M, Bioos S, Rahimi R, Malekshahi F, Nejatbakhsh F. Therapeutic efficacy of rose oil: A comprehensive review of clinical evidence. Avicenna J Phytomed. 2017 May-Jun;7(3):206-213. PMID 28748167

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03377088/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03377088/ICF_001.pdf